CLINICAL TRIAL: NCT00220623
Title: Efficacy and Cost-Effectiveness of 18-Months of Antidepressive Medication Plus Either Cognitive-Behavior Therapy or Dynamic Psychotherapy Compared to Supportive Clinical Management for Recurrent Major Depression: a Pilot Study
Brief Title: Efficacy of 18-Months of Antidepressive Medication Plus CBT or Dynamic or Supportive Psychotherapy for Recurrent Major Depression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #04-013
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Major Depression
Keywords: major depression; psychotherapy; antidepressant medications; clincial trial
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: antidepressant medications, flexible drug choice
Behavioral: CBT, Psychodynamic or Supportive Psychotherapy

SUMMARY:
Major Depressive Disorder affects approximately 16% of the adult population over the lifetime. Controlled studies indicate that short-term antidepressive medications or psychotherapy produce full remission in only about 46% of patients. Furthermore, about 80% of patients will continue to have subsequent recurrences after remission of the first episode, with each episode increasing the probability of future recurrences. This pilot study will examine whether antidepressive medications plus one of three commonly available types of psychotherapy used in the short-term treatment of depression can protect against the recurrence of depression if active treatment is extended to 18-months duration. Results will aid designing a more complete study.

Adults with an acute episode of major depressive disorder with at least one prior episode will be randomized to Antidepressive medications (ADM) plus 18-months of either Cognitive-behavioral therapy (CBT) or Dynamic psychotherapy (DYN), or to a standard control therapy, Supportive Clinical Management (SUP-CM). We will determine whether a higher percentage of those receiving either CBT or DYN remain well after three years of follow-up, compared to those receiving the standard control treatment. We will also examine the reduction in psychological risk factors as well as potential economic benefits of the three approaches.

DETAILED DESCRIPTION:
Major Depressive Disorder affects approximately 15% of the adult population over a lifetime. Controlled studies indicate that short-term antidepressive medications or psychotherapy produce full remission in only about 46% of patients. Furthermore, about 80% of patients will continue to have subsequent recurrences after remission of the first episode, with each episode increasing the probability of future recurrences. The World Health Organization estimates that by the year 2020 depression will be the second largest cause of medical disability worldwide. As a result, there is a need to validate treatments that produce remission and prevent recurrences upon long-term follow-up. Furthermore, since several treatment types are currently widely practiced, there is a need to demonstrate both their efficacies and cost effectiveness.

We propose to conduct a pilot study to determine the feasibility and provide estimates for a randomized controlled study of combined antidepressive medications plus one of three forms of psychotherapy in common use for adults with an acute episode of recurrent major depression. Two treatments of interest, Cognitive-behavioural (CBT) and psychodynamic (DYN) psychotherpy, will be compared to Supportive Clinical Management (SUP-CM), which will serve as the control. Overall, the study will compare each active psychotherapy to the control treatment for retention-attrition, and efficacy in producing remission, preventing recurrence after up to 18-months of treatment, and improving functioning. Secondary aims will explore whether putative psychological risk factors for depression improve more in the active psychotherapies than in the control condition, and determine whether this improvement predicts or mediates staying well. Finally, we will develop preliminary estimates of the cost-effectiveness and cost-offset of the three treatment conditions at termination and 3 year post-treatment follow-up. If either or both active treatments give estimates of superior prevention of recurrences or residual symptoms and impairment, these estimates will be used to plan a subsequent more definitive study, including their relative cost-effectiveness and cost-offset.

Adults (N=30, 10 per condition) meeting DSM-IV-TR criteria for an acute episode of major depressive disorder with at least one prior episode will be randomized to 18-months of either (1) Cognitive-behavioral therapy (CBT) or (2) Psychodynamic psychotherapy (DYN), to a standard control treatment (3) Supportive Clinical Management. All patients will receive antidepressive medications (ADM), which will be prescribed according to a pre-defined protocol similar to the CANMAT guidelines. Once remission has been achieved, continuation of ADM will follow the same guidelines in all three therapy conditions. Assessments will include the LIFE-method to code the course of depressive episodes and dysthymia, the HRSD-17 and BDI-2, role functioning and impulse symptom measures, and theoretically based measures of both cognitive, affective and dynamic psychological risk factors, and health care costs and economic productivity. Patients will be assessed at intake and six month intervals for the treatment period and three year subsequent follow-up, totaling up to 54 months for each patient. The HRSD-17 and economic data will be collected more frequently. Intent-to-treat analyses will compare each active treatment to the control treatment. If 18-months of either of these two most commonly used psychotherapies provides estimates of reduced recurrence and morbidity compared to standard treatment, these estimates will be used to design and power a subsequent complete study including cost-effectiveness and cost-offset.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV major depressive episode with at least one prior MDE episode, and
* HRSD-17 score above 16 at screening and intake (one-week apart)

Exclusion Criteria:

* bipolar type I disorder
* any psychotic disorder
* serious alcohol or substance abuse disorder
* organic mental disorder
* serious suicidal intent that warrants imminent hospitalization
* first trimester pregnancy
* likelihood of moving too far away to continue treatment for 18-months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-08

PRIMARY OUTCOMES:
Time to recovery of major depressive episode
Time to recurrence of major depression, once recovered
improvement in depressive defenses

SECONDARY OUTCOMES:
proportion of time with depressive symptoms
improvement on other specified psychological measures related to depression
cost-effectiveness measures

CONTACTS AND LOCATIONS:
Overall Officials: John C Perry, M.P.H., M.D., Principal Investigator — S.M.B.D. - Jewish General Hospital
Locations (1):
- Institute of Community and Family Psychiatry, Montreal, Quebec, Canada

REFERENCES:
- [Background] Trijsburg RW, Semeniuk TT, Perry JC. An Empirical Study of the Differences in Interventions between Dynamic Psychotherapy and Cognitive-Behavioral Therapy for Recurrent Major Depression. Canadian J Psychoanalysis 12(2): 325-345, 2004.